CLINICAL TRIAL: NCT04004208
Title: Open-label, Randomized, Two-Arm, Controlled Study to Assess the Efficacy, Safety, and Tolerability of Intravitreal (IVT) Aflibercept Compared to Laser Photocoagulation in Patients With Retinopathy of Prematurity (ROP)
Brief Title: Aflibercept for Retinopathy of Prematurity - Intravitreal Injection Versus Laser Therapy
Acronym: FIREFLEYE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20090; 2018-002611-99 (EudraCT Number)
Record Dates: First submitted 2019-06-28; First posted 2019-07-01 (Actual); Results first posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Retinopathy of Prematurity (ROP)
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aflibercept arm (Experimental): Subjects randomized to aflibercept will receive a intravitreal (IVT) injection of Dose A aflibercept per eligible eye at baseline and, if needed, up to a defined number of additional injections in each eye.
  Interventions: Drug: Eylea (Aflibercept, BAY86-5321)
- Laser photocoagulation arm (Active Comparator): Subjects randomized to laser photocoagulation will receive treatment in each eligible eye at baseline. Retreatments may be administered if needed.
  Interventions: Procedure: Laser photocoagulation

INTERVENTIONS:
Drug: Eylea (Aflibercept, BAY86-5321) — Solution in a sterile glass vial, Dose A, IVT injection.
  Arms: Aflibercept arm
Procedure: Laser photocoagulation — Transpupillary conventional laser ablative therapy
  Arms: Laser photocoagulation arm

SUMMARY:
The purpose of this study is to demonstrate how well aflibercept works in babies with ROP, comparing it with laser therapy. The study also has the objective to demonstrate how safe aflibercept is when used in babies, and describe how the drug moves into, through and out of the body.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth ≤ 32 weeks or birth weight ≤ 1500 g
* Subjects with treatment-naïve ROP classified according to the International Classification for ROP in at least one eye as:

  * Zone I Stage 1 plus, or 2 plus, or 3 non-plus or 3 plus, or
  * Zone II Stage 2 plus or 3 plus, or
  * Aggressive posterior retinopathy of prematurity (AP-ROP)
* Weight at baseline (day of treatment) ≥ 800 g
* Signed informed consent from parent(s)/legally authorized representative(s), which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Known or suspected chromosomal abnormality, genetic disorder or syndrome
* Previous exposure to any IVT or systemic anti-vascular endothelial growth factor (VEGF) agent, including maternal exposure during pregnancy and/or during breastfeeding
* Clinically significant neurological disease (eg, intraventricular hemorrhage grade 3 or higher, periventricular leukomalacia, congenital brain lesions significantly impairing optic nerve function, severe hydrocephalus with significantly increased intracranial pressure)
* Pediatric conditions rendering the infant ineligible for study intervention at baseline or for repeated blood draws as evaluated by a NICU specialist and a study ophthalmologist
* Presence of active ocular infection within 5 days of the first treatment
* Advanced stages of ROP with partial or complete retinal detachment (ROP Stages 4 and 5)
* ROP involving only Zone III
* Ocular abnormalities that may interfere with the administration of study intervention or assessment of the study primary endpoint
* Postnatal treatment with oral or intravenous corticosteroids at an equivalent dose of prednisone ≥ 1 mg/kg/day for > 2 weeks within 14 days of the first study intervention
* Previous surgical or nonsurgical treatment for ROP (IVT anti-VEGF injection, ablative laser therapy, cryotherapy, and vitrectomy)
* Participation of the subject or the mother in other clinical trials requiring administration of investigational treatments (other than vitamins and minerals) at the time of screening, or within 30 days or 5 half-lives of administration of the previous study drug, whichever is longer

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- Argentina (2):
  - Many Locations, Multiple Locations
  - Hospital Público Descentralizado "Dr. Guillermo Rawson", San Juan
- Austria (2):
  - Kepler Universitätsklinikum Campus III, Linz
  - Many Locations, Multiple Locations
- Belgium (2):
  - AZ St-Jan Brugge Oostende AV, Bruges
  - Many Locations, Multiple Locations
- Brazil (3):
  - Hospital das Clínicas de Botucatu - UNESP Botucatu, Botucatu, São Paulo
  - Many Locations, Multiple Locations
  - Unifesp/Epm, São Paulo
- Bulgaria (5):
  - Many Locations, Multiple Locations
  - UMHAT Sveti Georgi, Plovdiv
  - Acibadem City Clinic Multiprofile Hospital for Active Treatm, Sofia
  - II SOGHAT Sheinovo, Sofia
  - SHOGAT Prof Dimitar Stamatov, Varna
- Czechia (3):
  - Many Locations, Multiple Locations
  - Fakultni nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
- Greece (4):
  - P & A KYRIAKOU Children's Hospital, Athens
  - University General Hospital of Ioannina, Ioannina
  - Many Locations, Multiple Locations
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Many Locations, Multiple Locations
- Hungary (2):
  - EKBC, Uj Szent Janos Korhaz es Szakrendelo, Budapest
  - Many Locations, Multiple Locations
- Israel (2):
  - Many Locations, Multiple Locations
  - Kaplan Medical Center, Rehovot
- Italy (5):
  - IRCCS Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - A.O. di Perugia, Perugia, Umbria
  - Many Locations, Multiple Locations
- Japan (12):
  - University of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Okinawa Prefectural Nanbu Medical Center and Children's MC, Shimajiri-gun, Okinawa
  - Tokyo Metropolitan Children's Medical Center, Fuchū, Tokyo
  - Showa University Hospital, Shinagawa, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, Sumida-ku, Tokyo
  - Tokyo Metropolitan Ohtsuka Hospital, Toshima-ku, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Many Locations, Multiple Locations
  - Saitama Children's Medical Center, Saitama
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Many Locations, Multiple Locations
- Netherlands (2):
  - Many Locations, Multiple Locations
  - Maxima Medisch Centrum, locatie Veldhoven, Veldhoven
- Poland (2):
  - Many Locations, Multiple Locations
  - Ginekologiczno-Polozniczy SK UM im. K. Marcinkowskiego, Poznan
- Portugal (3):
  - Hospital Prof. Dr. Fernando Fonseca, Amadora, Lisbon District
  - CHLO - Hospital Sao Francisco Xavier, Lisbon
  - Many Locations, Multiple Locations
- Romania (3):
  - Clinical Emergency County Hospital, Cluj-Napoca, Cluj
  - Spitalul Clinic de Obstretica si Ginecologie "Cuza Voda", Iași
  - Many Locations, Multiple Locations
- Russia (6):
  - FSAI NMRC IRTC "Eye Microsurgery", Kaluga's Branch, Kaluga
  - Russian National Scientific Medical University, Moscow
  - FGBUZ "NPC of special children care n.a. Voino-Yaseneckogo", Moscow
  - Many Locations, Multiple Locations
  - Pediatric Medical University, Saint Petersburg
  - City Children Hospital ¿1, Saint Petersburg
- Singapore (2):
  - Many Locations, Multiple Locations
  - KK Women's and Children's Hospital, Singapore
- Slovakia (2):
  - Narodny ustav detskych chorob, Bratislava
  - Many Locations, Multiple Locations
- South Korea (4):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan-si, Chungcheongnam-do
  - Many Locations, Multiple Locations
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario "La Paz", Madrid
  - Hospital Regional de Málaga, Málaga
  - Many Locations, Multiple Locations
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Many Locations, Multiple Locations
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Many Locations, Multiple Locations
  - Mackay Memorial Hospital, Taipei
- Turkey (Türkiye) (7):
  - S.B.U. Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Baskent Universitesi Tip Fakultesi Hastanesi, Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Saglik Bilimleri Universitesi Antalya EA Hastanesi, Antalya
  - Eskisehir Osmangazi Universitesi Tip Fakultesi, Eskişehir
  - Many Locations, Multiple Locations
- Ukraine (2):
  - Many Locations, Multiple Locations
  - MI"Odesa Regional Children's Clinical Hospital", Odesa
- United Kingdom (2):
  - Birmingham Womens Hospital, Birmingham
  - Many Locations, Multiple Locations

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Stahl A, Azuma N, Wu WC, Lepore D, Sukgen E, Nakanishi H, Mazela J, Leal S, Pieper A, Schlief S, Eissing T, Turner KC, Zhao A, Winkler J, Hochel J, Kofuncu E, Zimmermann T; FIREFLEYE Study Group. Systemic exposure to aflibercept after intravitreal injection in premature neonates with retinopathy of prematurity: results from the FIREFLEYE randomized phase 3 study. Eye (Lond). 2024 Jun;38(8):1444-1453. doi: 10.1038/s41433-023-02919-9. Epub 2024 Jan 10. PMID 38200320
- [Derived] Stahl A, Sukgen EA, Wu WC, Lepore D, Nakanishi H, Mazela J, Moshfeghi DM, Vitti R, Athanikar A, Chu K, Iveli P, Zhao F, Schmelter T, Leal S, Kofuncu E, Azuma N; FIREFLEYE Study Group. Effect of Intravitreal Aflibercept vs Laser Photocoagulation on Treatment Success of Retinopathy of Prematurity: The FIREFLEYE Randomized Clinical Trial. JAMA. 2022 Jul 26;328(4):348-359. doi: 10.1001/jama.2022.10564. PMID 35881122
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 64 centers in 27 countries or regions, between 25-SEP-2019 (first participant first visit) and 12-Feb-2021 (last participant last visit).
Pre-assignment Details: 121 participants were screened. 1 participant was a screen fail and 2 participants were withdrawn by parent/guardian. 118 participants were randomized, 75 participants were randomized to the aflibercept arm and 43 to the laser arm. 113 participants were treated, 5 participants randomized to the laser photocoagulation arm were withdrawn before receiving any study intervention.
Groups:
- Aflibercept 0.4 mg: One intravitreal injection of aflibercept 0.4 mg (0.01 mL) per eligible eye at baseline (treatment), with up to 2 re-injections at the same single dose allowed for each eligible eye if required and interval since last aflibercept injection was 28 or more days. One or both eyes could be treated.
- Laser Photocoagulation: Laser treatment to each eligible eye at baseline (treatment), with supplementary laser treatments allowed. Multiple sessions within one week from baseline were counted as a single treatment. One or both eyes could be treated.
Period: Overall Study
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Started (All randomized participants who received any study treatment and had a baseline and at least one post-baseline assessment of efficacy (FAS)) | 75 | 38
SAF (The safety analysis set (SAF) included all participants who received any type of study treatment.) | 75 | 38
PKS (The pharmacokinetic analysis set (PKS) included all participants who received aflibercept treatment at the baseline visit and who had at least one nonmissing PK assessment following the first dose of study drug.) | 75 | 0
AAS (The anti-drug antibody (ADA) analysis set (AAS) included all participants who received aflibercept at baseline and had at least 1 nonmissing result in the ADA assay following the first study dose.) | 75 | 0
Completed | 68 | 36
Not Completed | 7 | 2
Not completed — Withdrawal by parent/guardian | 1 | 1
Not completed — Death | 3 | 0
Not completed — COVID-19 pandemic | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: SAF
Groups:
- Total: Total of all reporting groups
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation | Total
Number analyzed (Participants) | 75 | 38 | 113
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age at birth
  weeks | 26.43 (2.1) | 26 (1.6) | 26.29 (1.9)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 75 | 38 | 113
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 19 | 53
  Male | 41 | 19 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 55 | 28 | 83
  Black or African American | 2 | 0 | 2
  Asian Indian | 0 | 2 | 2
  Chinese | 4 | 0 | 4
  Japanese | 10 | 6 | 16
  Korean | 2 | 1 | 3
  Asian: Other | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 1 | 1
  Multiple | 1 | 0 | 1
ROP classification by investigator [Count of Participants; unit: Participants] — ROP (retinopathy of prematurity) classified by the investigator according to the International Classification for Retinopathy of Prematurity in at least one eye with one of the following retinal findings: Zone I, or Zone II, or AP(aggressive posterior)-ROP (Zone I, Zone II). Zone I is the innermost zone of the retina centered around the optic disc, surrounded by the more peripheral Zone II. AP-ROP is a rapidly progressive form of ROP, with posterior location, most commonly observed in Zone I, less common in posterior Zone II. AP-ROP, if untreated, usually progresses to retinal detachment.
  Participants
    Zone I excluding AP-ROP | 15 | 7 | 22
    Zone II excluding AP-ROP | 46 | 26 | 72
    AP-ROP: Zone I | 12 | 4 | 16
    AP-ROP: Zone II | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Absence of Active ROP and Unfavorable Structural Outcomes
Description: Active ROP was defined as ROP requiring treatment. Unfavorable structural outcomes included retinal detachment, macular dragging, macular fold, or retrolental opacity.
Time Frame: At 24 weeks after starting study treatment
Measure: Number; unit: Proportion of participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Proportion of participants | 0.855 | 0.821
Statistical Analysis 1: Comparison: Aflibercept 0.4 mg vs Laser Photocoagulation; Bayesian analysis with non-informative prior distributions. Calculation of two-sided 90% credible interval for the treatment difference (aflibercept - laser photocoagulation); Test type: Non-Inferiority — Non inferiority margin is 5%. Confidence interval actually refers to a credible interval based on the Bayesian analysis; Difference in proportions = 0.034, 90% CI 2-sided [-0.08 to 0.162]

2. Secondary Outcome: Proportion of Participants Requiring Intervention With a Second Treatment Modality
Description: A second treatment modality for ROP was either rescue treatment or any other surgical or nonsurgical treatment for ROP (e.g. IVT anti-VEGF injection, ablative laser therapy, cryotherapy, or vitrectomy) captured as concomitant medication or surgery after study start.
Time Frame: From baseline (treatment) up to week 24.
Measure: Number; unit: Proportion of participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Proportion of participants | 0.072 | 0.096
Statistical Analysis 1: Comparison: Aflibercept 0.4 mg vs Laser Photocoagulation; [analysis description as in outcome 1, analysis 1]; Test type: Other — Confidence interval actually refers to a credible interval based on the Bayesian analysis; Difference in proportions = -0.023, 90% CI 2-sided [-0.11 to 0.046]

3. Secondary Outcome: Proportion of Participants With Recurrence of ROP
Description: Participants with recurrence of ROP were defined as subjects requiring re-treatment or rescue treatment after in the past the absence of treatment-requiring active ROP had been confirmed by the investigator.
Time Frame: From baseline (treatment) up to week 24.
Measure: Number; unit: Proportion of participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Proportion of participants | 0.161 | 0.063
Statistical Analysis 1: Comparison: Aflibercept 0.4 mg vs Laser Photocoagulation; [analysis description as in outcome 1, analysis 1]; Test type: Other — Confidence interval actually refers to a credible interval based on the Bayesian analysis; Difference in proportions = 0.096, 90% CI 2-sided [0.019 to 0.175]

4. Secondary Outcome: Exploration of ROP Activity Scale Proposed by the International Neonatal Consortium
Description: Eyes were evaluated for change in ROP activity scale proposed by the International Neonatal Consortium (2018). ROP Activity Scale value range is from 0 to 22. Value 0 to 7 are considered mild, 8 to 12 are moderate, and 13 to 22 are severe. Value 0 means the best and value 22 means the worst. Eyes evaluation was done at baseline and each visit.
Time Frame: From baseline (treatment) up to week 24.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Scores on a scale
  Baseline | 16.20 (2.81) [lower limit 2.81] | 15.63 (3.53) [lower limit 3.53]
  Change from baseline to Week 24 | -15.42 (4.46) [lower limit 4.46] | -14.77 (4.19) [lower limit 4.19]

5. Secondary Outcome: Percentage of Participants With Ocular Treatment-emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that was observed or reported after the first and not later than 30 days after the last administration of study treatment. Participants treated after week 21 were followed-up for adverse events up to week 28. Ocular TEAEs in treated eyes only were reported
Time Frame: From baseline (treatment) up to week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Percentage of participants | 38.7 | 36.8

6. Secondary Outcome: Percentage of Participants With Ocular Serious Adverse Events (SAEs)
Description: Participants treated after week 21 were followed-up for adverse events up to week 28. Ocular SAEs in treated eyes only were reported.
Time Frame: From baseline (treatment) up to week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Percentage of participants | 13.3 | 7.9

7. Secondary Outcome: Percentage of Participants With Systemic TEAEs
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that was observed or reported after the first and not later than 30 days after the last administration of study treatment. Participants treated after week 21 were followed-up for adverse events up to week 28. Systemic TEAEs only were reported.
Time Frame: From baseline (treatment) up to week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Percentage of participants | 52.0 | 63.2

8. Secondary Outcome: Percentage of Participants With Systemic SAEs
Description: Participants treated after week 21 were followed-up for adverse events up to week 28. Systemic SAEs only were reported.
Time Frame: From baseline (treatment) up to week 24
Measure: Number; unit: Percentage of participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Percentage of participants | 24.0 | 36.8

9. Secondary Outcome: Concentrations of Free Aflibercept in Plasma
Description: Blood samples for determination of aflibercept concentrations in plasma were collected in the aflibercept 0.4 mg arm at Day 1 (within 24 hours after injection), and at weeks 2 and 4, and if feasible also at weeks 8, 12 and 24. Statistics for week 8, 12, 24 not calculated as > 1/3 of the concentrations were below the lower limit of quantification. Free Aflibercept Concentrations in Plasma were only measured in the Aflibercept 0.4 mg treatment arm.
Time Frame: From Day 1 up to week 24.
Population: The outcome measure was analyzed based on pharmacokinetic analysis set (PKS). The PKS included all participants who received aflibercept treatment at the baseline visit and who had at least one nonmissing PK assessment following the first dose of study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Aflibercept 0.4 mg
Number analyzed (Participants) | 75
ng/mL
  WEEK 0, DAY 1 | 480.607 (884.724)
  WEEK 2: number analyzed (Participants) | 66
  WEEK 2 | 218.965 (358.933)
  WEEK 4: number analyzed (Participants) | 68
  WEEK 4 | 133.093 (205.052)

10. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA)
Description: Immunogenicity was characterized by anti-drug antibody (ADA) responses in patients in the aflibercept 0.4 mg arm. Serum samples were taken at baseline prior to the injection and at 12 weeks after injection. ADA titers were summarized for 3 categories: Low (titer <1,000); Moderate (1,000 ≤ titer ≤ 10,000); High (titer >10,000). ADA in serum were only measured in the Aflibercept 0.4 mg treatment arm.
Time Frame: Baseline (treatment) and 12 weeks after aflibercept injection
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 0.4 mg
Number analyzed (Participants) | 75
Participants
  Baseline: ADA positive response | 0
  Baseline: ADA negative response | 75
  Week 12: ADA positive response | 1
  Week 12: ADA negative response | 74

11. Secondary Outcome: Number of Participants With Potential Neutralizing Antibodies (NAb)
Description: NAb status was evaluated for the samples that were positive in the ADA assay and had sufficient volume to analyze. NAb were only measured in participants with positive ADA in the Aflibercept 0.4 mg treatment arm
Time Frame: At 12 weeks after aflibercept injection
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 0.4 mg
Number analyzed (Participants) | 1
Participants | 0

12. Secondary Outcome: Number of Aflibercept Administrations
Description: Total number of injections in both eyes.
Time Frame: From baseline (treatment) up to week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Participants
  0 aflibercept administration | 0 | 34
  1 aflibercept administration | 4 | 0
  2 aflibercept administrations | 55 | 3
  3 aflibercept administrations | 6 | 1
  4 aflibercept administrations | 10 | 0

13. Secondary Outcome: Number of Laser Treatments
Description: Total number of laser treatment in both eyes. If multiple sessions of laser treatment were necessary within 1 week from baseline, they were counted as a single treatment.
Time Frame: From baseline (treatment) up to week 24.
Measure: Count of Participants; unit: Participants
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
Number analyzed (Participants) | 75 | 38
Participants
  0 laser treatment | 70 | 0
  1 laser treatment | 3 | 4
  2 laser treatments | 2 | 30
  3 laser treatments | 0 | 1
  4 laser treatments | 0 | 2
  6 laser treatments | 0 | 1

ADVERSE EVENTS:
Time Frame: After the first administration and not later than 30 days after the last administration of study treatment, up to 24 weeks.
Description: Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study.
Arm/Group | Aflibercept 0.4 mg | Laser Photocoagulation
All-Cause Mortality (participants affected / at risk) | 3/75 | 0/38
Serious Adverse Events (participants affected / at risk) | 9/75 | 10/38
Other Adverse Events (participants affected / at risk) | 53/75 | 23/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 0.4 mg (N=75) | Laser Photocoagulation (N=38)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Corneal oedema (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 3 (3) | 2 (2)
Retinal haemorrhage (Eye disorders) | 2 (2) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infantile apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept 0.4 mg (N=75) | Laser Photocoagulation (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Anaemia neonatal (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital arterial malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Auditory disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1) | 0 (0)
Adrenomegaly (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 4 (6) | 0 (0)
Conjunctival oedema (Eye disorders) | 2 (4) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 1 (2)
Eyelid oedema (Eye disorders) | 2 (4) | 3 (5)
Iris adhesions (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (2) | 0 (0)
Lenticular opacities (Eye disorders) | 1 (2) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 0 (0)
Retinal haemorrhage (Eye disorders) | 4 (7) | 5 (6)
Retinal vascular disorder (Eye disorders) | 1 (2) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 2 (3) | 1 (2)
Swelling of eyelid (Eye disorders) | 1 (2) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vitreous opacities (Eye disorders) | 1 (2) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 1 (2) | 0 (0)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crying (General disorders) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 3 (3) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 2 (2)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (5) | 3 (5)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Multiple use of single-use product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Intraocular pressure increased (Investigations) | 2 (3) | 0 (0)
Oxygen saturation decreased (Investigations) | 3 (4) | 0 (0)
Brain stem auditory evoked response abnormal (Investigations) | 2 (3) | 0 (0)
Otoacoustic emissions test abnormal (Investigations) | 2 (3) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Developmental coordination disorder (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 1 (1) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Neonatal seizure (Nervous system disorders) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction is that the PI has to ensure that the sponsor can review results communications at least 60 days prior to the planned public release.

DOCUMENTS (2):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT04004208/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT04004208/SAP_001.pdf